CLINICAL TRIAL: NCT04328064
Title: The Role of Rosuvastatin on Vascular Involvement in Behçet's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Professor of Rheumatology, University of Alexandria
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alexmed116619312
Record Dates: First submitted 2011-08-29; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Behcet's Disease
Keywords: Behcet's Disease; Rosuvastatin; Vascular Markers; Improvement in vascular involvement in Behcet's Disease
MeSH Terms: conditions — Behcet Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin Drug (Active Comparator): Active drug-rosuvastatin 40 mg
  Interventions: Drug: Rosuvastatin calcium 40mg; Drug: Placebo oral tablet
- Placebo drug (Placebo Comparator): Placebo oral tablet
  Interventions: Drug: Rosuvastatin calcium 40mg; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Rosuvastatin calcium 40mg — Active drug -Rosuvastatin
  Other Names: Experimental active drug
Drug: Placebo oral tablet — 40 mg placebo for 12 months
  Other Names: Placebo comparator

SUMMARY:
Behçet's Disease(BD) is a systemic inflammatory vasculitis, which affects all types and sizes of vessels. Statins display numerous effects often independent of the well-established lipid-lowering effects that may be of benefit in retarding or preventing vascular injury and ischaemic vascular events. The aim of the present study was to determine the efficacy of rosuvastatin in improving vascular dysfunction and vascular inflammation and to assess the effect of rosuvastatin on vascular involvement in BD patients. Fifty-six BD patients (51 males and 5 females) mean age 33.4 years, mean disease duration 5.8 years), all fulfilling the classification criteria of the International Study Group for Behçet's disease were recruited.Patients were randomised into 2 groups.

The first group (n=27: 20 active and 7 inactive) were assigned to receive 40 mg of rosuvastatin and the second group(n=29: 21 active and 8 inactive) received placebo for 12 months. Inflammatory and endothelial dysregulation markers were measured at baseline and after 12 months. All patients were examined for vascular involvement. Venous or arterial system involvement was defined as present when confirmed by Doppler ultrasonography, magnetic resonance angiography, conventional angiography or CT.

ELIGIBILITY:
Inclusion Criteria:

* all patients fulfilling the classification criteria of the International Study Group for Behçet's disease

Exclusion Criteria:

* smoking,
* diabetes mellitus,
* hypercholesterolaemia,
* hypertension,
* cardiac insufficiency,
* coexisting hepatic and renal diseases
* inflammatory diseases.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial and vascular inflammatory markers | 12 months
  Outcome measures included alterations in endothelial injury and vascular inflammatory markers.

SECONDARY OUTCOMES:
Occurrence of new-onset vascular involvement | 6 months